CLINICAL TRIAL: NCT07108387
Title: A Randomized Study of Tocilizumab Discontinuation for Patients With Giant Cell Arteritis in Remission (AGA01)
Brief Title: Tocilizumab Discontinuation Versus Dose Reduction for Patients With Well-Controlled Giant Cell Arteritis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DAIT AGA01
Record Dates: First submitted 2025-07-18; First posted 2025-08-07 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Giant Cell Arteritis (GCA)
Keywords: Tocilizumab; Giant Cell Arteritis; ACTEMRA(R)
MeSH Terms: conditions — Giant Cell Arteritis | interventions — tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tocilizumab Step-Down Dosing Arm (Experimental): Randomization will be performed within strata defined by gender, whether the participant has a history of Giant cell arteritis (GCA) relapse, and whether the participant has a history of polymyalgia rheumatica (PMR) symptoms.
  Patients in remission of high dose Tocilizumab (TCZ) >=12months and discontinued glucocorticoids (e.g. prednisone) >=3 months will receive 162mg subcutaneously (SC) every 2 weeks or 4mg/Kg intravenously (IV) monthly for 18 months
  Participants who remain in remission will enter the Follow-Up Phase for an additional 12 months at Month 18 and will discontinue TCZ at that time
  Interventions: Drug: Tocilizumab
- Tocilizumab Withdrawal Arm (Other): Randomization will be performed within strata defined by gender, whether the participant has a history of Giant cell arteritis (GCA) relapse, and whether the participant has a history of PMR symptoms.
  Patients in remission of high dose Tocilizumab (TCZ) >=12months and discontinued glucocorticoids (e.g. prednisone) >=3 months will discontinue Tocilizumab and will have visits at Week 2, Month 1 and 2, and then every 2 months during the TCZ Withdrawal Phase until the Month 18 Visit.
  Participants who remain in remission will enter the Follow-Up Phase for an additional 12 months at Month 18 and will continue withdrawal at that time.
  Interventions: Drug: Discontinue Tocilizumab

INTERVENTIONS:
Drug: Tocilizumab — Participants will continue Tocilizumab (TCZ) at a lower dose of either 4 mg/kg IV monthly or 162 mg SC every 2 weeks
  Participants randomized to the stepped-down treatment arm will receive TCZ on their current route of administration. The route of administration may change if needed during study participation at the discretion of the investigator
  Other Names: ACTEMRA
  Arms: Tocilizumab Step-Down Dosing Arm
Drug: Discontinue Tocilizumab — Participants will discontinue Tocilizumab and will have visits at Week 2, Month 1 and 2, and then every 2 months during the TCZ Withdrawal Phase until the Month 18 Visit.
  Participants who remain in remission will enter the Follow-Up Phase for an additional 12 months at Month 18 and will continue withdrawal at that time.
  Other Names: ACTEMRA
  Arms: Tocilizumab Withdrawal Arm

SUMMARY:
This is a multi-center, randomized, open label study that will assess the efficacy and safety of ACTEMRA(R) or one of its FDA-approved biosimilars Tocilizumab (TCZ) maintenance versus withdrawal in Giant cell arteritis (GCA) patients who are in remission after at least 12 months of high dose TCZ treatment. Eligible participants will also have discontinued glucocorticoids (e.g., prednisone (or equivalent)) entirely at least three months before randomization. High dose TCZ treatment includes 6-8 mg/kg intravenously (IV) monthly or 162 mg subcutaneously (SC) weekly, which are two forms of administration that are commonly used in clinical practice and are equally efficacious in controlling GCA

This research study has three parts:

1. The screening phase (up to 42 days) consists of collecting information about your health and your GCA, a physical exam, and blood tests to see If you qualify to enroll in the study
2. The study treatment phase (withdrawal/step down dosing phase study months 0 - 18) consists of you either completely stopping or decreasing your current dose of tocilizumab while collecting information about your health and your GCA as well as blood samples every two months at clinic visits
3. The safety follow-up phase (months 19-30) consists of collecting information about your health and your GCA as well as blood samples every three months

The primary objective is to determine the rate of disease relapse at 18 months in participants with GCA who receive low-dose TCZ compared to those who discontinue TCZ

ELIGIBILITY:
Inclusion Criteria:

1. Ability and willingness to provide written informed consent and to comply with the study protocol
2. Diagnosis of Giant cell arteritis (GCA) classified according to the following criteria:

   a. AND at least one of the following:

   i. Cranial signs or symptoms of GCA (new-onset localized headache, scalp tenderness, temporal artery tenderness or decreased pulsation, ischemia-related vision loss, or otherwise unexplained mouth or jaw pain upon mastication)

   ii. Symptoms of polymyalgia rheumatica (PMR), defined as shoulder and / or hip girdle pain associated with inflammatory morning stiffness

   b. AND at least one of the following:

   i. Artery biopsy revealing features of GCA (e.g., mononuclear cell infiltration or granulomatous inflammation)

   ii. Evidence of large-vessel vasculitis by angiography or cross-sectional imaging study such as ultrasound (US), Magnetic resonance angiography (MRA), computerized tomography angiography (CTA), or Positron emission tomography-computerized tomography (PET-CT)

   iii. Ultrasound (US) or Magnetic resonance imaging (MRI) or PET/CT demonstration of features of GCA in a cranial artery
3. Glucocorticoid-free remission on Tacrolimus (TCZ) therapy according to the following criteria:

   1. Ongoing treatment with TCZ (ACTEMRA(R) or one of its FDA-approved biosimilars) administered at 6-8 mg/kg IV every 4 weeks OR 162 mg subcutaneous (SC) weekly for at least 12 months prior to randomization. Participants cannot have missed more than one SC dose or any Intravenously (IV) doses in the 2 months prior to randomization
   2. Disease remission for at least 12 months prior to randomization defined as the absence of clinical signs or symptoms of active GCA and Polymyalgia rheumatica (PMR) along with normal values of C-reactive protein (CRP) (< 10 mg/L) at screening
   3. Absence of oral, IV, intramuscular (IM), or SC glucocorticoid treatment for at least 3 months prior to randomization

Exclusion Criteria:

1. An autoimmune disease or other condition, other than Giant cell arteritis (GCA), that requires/is anticipated to require chronic or recurrent oral or parenteral glucocorticoids or other immunomodulatory therapy. (Topical and inhaled therapies are acceptable)
2. Hospitalization within 8 weeks prior to randomization
3. Suspected or established adrenal insufficiency
4. Treatment with any investigational agent within 12 months of randomization
5. Concomitant treatment with another biologic immunosuppressant (e.g., etanercept, adalimumab, infliximab, certolizumab, golimumab, sarilumab, abatacept, rituximab, or secukinumab) within 12 months prior to randomization. Concomitant treatment with non-biologic immunosuppressants (e.g.

   JAK inhibitors, Methotrexate (MTX)) within 3 months prior to randomization. An exception is hydroxychloroquine, which is permitted as long as the dose has been stable for the 8 weeks preceding randomization
6. Immunization with a live/attenuated vaccine within <= 4 weeks prior to randomization
7. History of severe allergic or anaphylactic reactions to Tocilizumab (TCZ) or to prednisone (or equivalent)
8. Evidence of serious uncontrolled concomitant cardiovascular, nervous system, pulmonary (including obstructive pulmonary disease), renal, hepatic, endocrine (including uncontrolled diabetes mellitus), psychiatric, osteoporosis/osteomalacia, glaucoma, corneal ulcers/injuries, or gastrointestinal (GI) disease
9. Serologic evidence of chronic hepatitis infection at time of TCZ initiation or at screening if not previously assessed:

   1. Evidence of current or prior infection with hepatitis B, as indicated by a positive test for the hepatitis B surface antigen or an isolated positive test for the hepatitis B core antibody. If a participant has an isolated positive hepatitis B core antibody, clearance after consultation with infectious disease specialist or gastroenterologist/hepatologist must be obtained
   2. Evidence of current or prior infection with hepatitis C virus (HCV), except adequately treated HCV with sustained virologic response >= 12 weeks. If a participant has a positive or indeterminate hepatitis C antibody, viral load testing (e.g., reflex testing) is required. Clearance after consultation with infectious disease specialist or gastroenterologist/hepatologist must be obtained
10. Positive interferon gamma release assay (IGRA) (e.g., QuantiFERON Gold or equivalent) at time of TCZ initiation or at screening if not previously assessed

    1. If the participant has had the BCG vaccine or has some other condition complicating the interpretation of tuberculosis (TB) testing, clearance after consultation with infectious disease specialist or pulmonologist must be obtained
    2. Participants diagnosed with latent TB are eligible but must have initiated appropriate prophylaxis for at least 30 days prior to initiation of study treatment
    3. Indeterminate IGRA must be repeated (with same or other IGRA per local policy) and shown to be negative. Alternatively, if the IGRA remains indeterminate, a participant must have a negative PPD
11. Known active bacterial, viral, fungal, mycobacterial, or other infections except fungal infections of the nail beds and superficial cutaneous infection treated topically
12. Participant is pregnant or breastfeeding or planning a pregnancy while enrolled in the study
13. Any infection requiring treatment with IV antibiotics within 4 weeks of randomization or oral antibiotics within 2 weeks of randomization
14. Active treatment for malignancy at the time of randomization, with exception of prophylactic hormonal therapy (e.g. prostate cancer, breast cancer, etc.)
15. History of alcohol, drug, or chemical abuse within 12 months prior to randomization
16. History of chronic or recurrent infection (excluding simple cystitis, viral respiratory infection, sinusitis, dermatophyte (tinea) infection) within 12 months prior to randomization
17. History of opportunistic infection within 12 months prior to randomization unless evaluated and cleared by an infectious disease or pulmonary specialist
18. Any of the following laboratory values during screening:

    1. Alanine Transaminase (ALT) or Aspartate Aminotransferase (AST) > 1.5 × upper limit of normal (ULN)
    2. Platelet count < 100 × 10^9/L (100,000/mm^3)
    3. Hemoglobin (Hb) < 90 g/L (9 g/dL; 5.6 mmol/L)
    4. White blood cells < 3.0 × 10^9/L (3000/mm^3)
    5. Absolute neutrophil count (ANC) < 1.0 × 10^9/L (1000/mm^3)
19. Past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements, or that may impact the quality or interpretation of the data obtained from the study

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2025-12-11 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients in sustained remission | Through Month 18
  Sustained remission and clinical relapse will be determined by the investigator based on clinical signs and symptoms of active Giant cell arteritis (GCA) and PMR regardless of the values of erythrocyte sedimentation rate (ESR) and C-reactive protein (CRP). The absence of clinical signs and symptoms of active GCA and PMR over the TCZ Withdrawal/Step-Down Dosing and Follow-Up Phases will define sustained remission through Months 18 and 30, respectively. Clinical relapse will be based on recurrent signs or symptoms attributed to GCA regardless of the values of ESR and CRP. To fulfill the definition of a disease relapse, the investigator must make the decision to intensify the participants GCA treatment

SECONDARY OUTCOMES:
Time to disease relapse | Through Month 30
Number of disease relapses | At Months 18 and 30
Annualized relapse rate | At Months 18 and 30
Cumulative prednisone (or equivalent) dose | At Months 18 and 30
Cumulative Glucocorticoid Toxicity Index (GTI) excluding the bone density domain | At Months 18 and 30
  calculated as the cumulative worsening score (CWS) and aggregate improvement score (AIS)
Clinical features of disease relapse | Through Month 30
  Sustained remission and clinical relapse will be determined by the investigator based on clinical signs and symptoms of active Giant cell arteritis (GCA) and PMR regardless of the values of ESR and CRP. The absence of clinical signs and symptoms of active GCA and PMR over the TCZ Withdrawal/Step-Down Dosing and Follow-Up Phases will define sustained remission through Months 18 and 30, respectively. Clinical relapse will be based on recurrent signs or symptoms attributed to GCA regardless of the values of ESR and CRP. To fulfill the definition of a disease relapse, the investigator must make the decision to intensify the participants GCA treatment
The number of Adverse Events (AEs) | At Months 18 and 30
The nature of Adverse Events (AEs) | At Months 18 and 30
The severity of Adverse Events (AEs) | At Months 18 and 30
The number of Serious Adverse Events (SAEs) | At Months 18 and 30
The nature of Serious Adverse Events (SAEs) | At Months 18 and 30
Proportion of patients in sustained remission | Through Month 30

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian H Unizony, M.D., Study Chair — Massachusetts General Hospital: Rheumatology, Allergy and Immunology, Center for Immunology and Inflammatory Diseases
Locations (7):
- United States (7):
  - Emory University School of Medicine: Division of Rheumatology, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Johns Hopkins Hospital: Division of Rheumatology Vasculitis Center, Baltimore, Maryland
  - Massachusetts General Hospital: Rheumatology, Allergy and Immunology, Center for Immunology and Inflammatory Diseases, Boston, Massachusetts
  - Northwell Health: Division of Rheumatology and Allergy-Clinical Immunology, Great Neck, New York
  - Hospital for Special Surgery, New York: Division of Rheumatology, New York, New York
  - University of Pittsburgh Medical Center: Division of Rheumatology and Clinical Immunology, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Immunology Database and Analysis Portal (ImmPort), a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts.
Time Frame: On average, within 24 months after database lock for the trial.
Access Criteria: Open access
URL: http://www.immport.org/home

REFERENCES:
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — http://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait